CLINICAL TRIAL: NCT00546507
Title: The Efficacy and Safety of TDS-943 in the Treatment of Osteoarthritis of the Knee: Pivotal Study I
Brief Title: Study Evaluating the Efficacy and Safety of Topical Diclofenac Spray in Osteoarthritis of the Knee: Trial I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mika Pharma GmbH (Industry)
Responsible Party: Bernd G. Seigfried, MIKA Pharma GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TD-06-13
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator): placebo
  Interventions: Other: placebo
- B (Active Comparator): celecoxib 200 mg qd p.o.
  Interventions: Drug: celecoxib
- C (Experimental): TDS-943 40 mg bid topically
  Interventions: Drug: TDS-943 (topical diclofenac sodium 4% spray)

INTERVENTIONS:
Drug: TDS-943 (topical diclofenac sodium 4% spray)
  Arms: C
Drug: celecoxib
  Arms: B
Other: placebo
  Arms: A

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of TDS-943 (topical diclofenac spray) compared to oral celecoxib and placebo in subjects with osteoarthritis of the knee. The main hypotheses are that TDS-943 will be better than placebo and no worse than celecoxib.

DETAILED DESCRIPTION:
This is a multicenter, outpatient, multiple-dose, placebo- and active controlled, double-blind, double-dummy parallel group, randomized (stratified by unilateral vs. bilateral knee OA) trial. The trial will enroll subjects who have been diagnosed with OA of the knee (confirmed by weight-bearing x-ray) and whose condition is in flare at baseline. Subjects who qualify to enter the study will be randomized to topical TDS-943 40 mg bid, oral celecoxib 200 mg qd, or placebo in a 3:2:2 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Males or females in generally good health at least 40 years of age
* Osteoarthritis (OA) of at least one knee, verified by a weight-bearing radiograph
* Subject has taken an oral NSAID or analgesic at least 3 days during the past 30 days to treat knee OA pain

Exclusion Criteria:

* Females who are pregnant or lactating or who may become pregnant
* Hypersensitivity (exacerbations of asthma, rhinitis, or urticaria) to sulfonamides, acetaminophen, diclofenac, celecoxib, aspirin, or any other NSAID
* History of myocardial infarction, congestive heart failure, stroke, coronary-artery bypass graft surgery, or any other significant cardiovascular disease, or is on any form of anticoagulation therapy other than low-dose aspirin (no more than 325 mg/day)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC Composite Pain Score | 30 days

SECONDARY OUTCOMES:
Change from baseline in the WOMAC Composite Stiffness and Composite Function Scores, Change from Baseline in the Subject's Global Assessment of Arthritic Condition, Change from baseline in the Subject's Assessment of OA Pain, %OMERACT-OARSI responders | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Mika Pharma GmbH
Locations (38):
- United States (38):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - Fair Oaks, California
  - Pico Rivera, California
  - Santa Barbara, California
  - Torrance, California
  - DeLand, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Gurnee, Illinois
  - Morton, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - Baton Rouge, Louisiana
  - Florissant, Missouri
  - St Louis, Missouri
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Perrysburg, Ohio
  - Wallingford, Pennsylvania
  - Cranston, Rhode Island
  - Cordova, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Roanoke, Virginia